CLINICAL TRIAL: NCT06531707
Title: Efficacy and Safety of Ibuprofen/Loratadine Fixed-dose Combination Versus the Fixed-dose Administration of Monotherapy as Symptomatic Treatment for Patients With the Common Cold
Brief Title: Efficacy and Safety in the Combination of Ibuprofen / Loratadine Versus Ibuprofen Versus Loratadine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30700-III-23(1)
Record Dates: First submitted 2024-07-18; First posted 2024-08-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Common Cold
Keywords: Common Cold; Flu; Ibuprofen; Loratadine
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — Ibuprofen; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen + Loratadine (Experimental): Administered orally (suspension), 5 mL twice a day, for 7 days.
  Interventions: Drug: Ibuprofen + Loratadine fixed dose
- Ibuprofen (Active Comparator): Administered orally (suspension), 20 mL, twice a day for 7 days.
  Interventions: Drug: Ibuprofen
- Loratadine (Active Comparator): Administered orally (suspension), 5 mL, twice a day for 7 days
  Interventions: Drug: Loratadine

INTERVENTIONS:
Drug: Ibuprofen + Loratadine fixed dose — Suspension 8,000 mg / 100 mg / 100 mL, 5 mL twice a day
  Other Names: Ibu+Lora
  Arms: Ibuprofen + Loratadine
Drug: Ibuprofen — Suspension 2,000 mg / 100 mL, 20 mL twice a day
  Other Names: Ibu
  Arms: Ibuprofen
Drug: Loratadine — Suspension 1 mg / 1 mL, 5 mL twice a day
  Other Names: Lora
  Arms: Loratadine

SUMMARY:
Phase III longitudinal, multicenter, randomized, double-blind clinical trial. The aim of this study is to evaluate the efficacy and safety of the drug combination of Ibuprofen/Loratadine versus Ibuprofen versus Loratadine as monotherapy for the symptomatic treatment of the common cold.

DETAILED DESCRIPTION:
Researchers will compare the fixed-dose combination of Ibuprofen + Loratadine versus Ibuprofen versus Loratadine for the symptomatic treatment of the common cold. The adverse events related to the interventions will be registered during follow up.

In the event that the symptoms worsen or the patient's clinical condition warrants the use of any additional medication, the principal investigator or designated physician will be in charge of prescribing it according to the individual clinical condition and the physical examination, this will be recorded as "Concomitant medication".

Participants will:

* Be randomized into one of the 3 intervention groups (A,B,C)
* Visit the clinic at day 0 (day of enrollment) and at day 7
* Answer the first symptomatic related survey at the randomization visit (V0) and the following ones in the morning when they wake up, the last survey will be answered at the final visit (day 7)

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study and give written informed consent
* At least 6 points on the Jackson scale according to physical examination and questioning (sneezing, runny nose, nasal obstruction, sore throat, cough, headache, malaise, and chills).
* Symptoms associated with the common cold with maximum of 3 days since presentation
* Women of childbearing potential under a medically acceptable method of contraception
* At the discretion of the Principal Investigator (PI) or treating physician, treatment with the researching product is indicated and may present clinical benefit

Exclusion Criteria:

* Patients in whom respiratory symptoms are suspected to be of bacterial origin and generate a clinical picture compatible with: Rhinosinusitis (muco-purulent discharge, headache or facial pain, etc.), lower respiratory tract disease (wheezing, crackles, productive cough, etc.), acute otitis media (otalgia, purulent discharge from the ear, auditory discomfort, etc.).
* Patients participating in another clinical trial involving an investigational treatment or participation in one within 4 weeks prior to study start
* Patients in whom participation in the study may be influenced (employment relationship with the research site or sponsor, inmates, etc.)
* At medical discretion, a disease that affects prognosis and prevents outpatient management, for example, but not limited to: end-stage cancer, kidney, heart, respiratory or liver failure, mental illness or with scheduled surgical or hospital procedures
* History/presence of any disease or condition that, in the opinion of the Investigator, could pose a risk for the patient or confusing the efficacy and safety of the investigational product
* Patients in whom the study drug is contraindicated for medical reasons
* Patients with allergy or hypersensitivity to the active substance of the study drugs, related products or excipients (Ibuprofen of Loratadine)
* Pregnant women, women breastfeeding or planning a pregnancy during the conducting the study
* Significant history of gastrointestinal diseases (e.g., gastric ulcer, Crohn's disease, Ulcerative Colitis, etc.)
* History of chronic liver failure Child-Pugh A, B, and/or C
* History of acute renal failure (glomerular filtration rate <30 ml/min/1.72 m2)
* Patients with a history of alcohol or drug abuse in the last year
* Patients with symptoms suggestive of COVID-19 infection (fever, cough, dyspnea) and/or contact in the last 14 days with a suspected or positive patient for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Assess the improvement in symptoms, comparing the percentage change through the Jackson score | 7 days
  The Jackson score is calculated by summing 8 symptom scores (sneezing, headache, malaise, chilliness, nasal discharge, nasal obstruction, sore throat and cough), rated as 0=absent, 1=mild, 2=moderate, and 3=severe.
Number of participants with treatment-related adverse events through the patient's diary record, by treatment group | 7 days
  To describe the frequency, intensity and causality of the adverse events presented during the clinical trial by treatment group. The adverse events will be registered by the patient in the diary record. Each adverse event will be followed up at the discretion of the researcher

SECONDARY OUTCOMES:
Assess the subjective change in patients in relation to quality of life through the modified Likert score | 7 days
  To compare quality of life measured as a difference in the modified Likert score by treatment group during the 7 days after starting treatment with respect to the baseline measurement. The patient will answer the scale daily.
  The Likert Scale is a seven point scale that is used to allow an individual to express how much they agree or disagree with a particular statement. The scale consists of 1 question associated to quality of life. The possible answers go from No interference to Severe interference.
Assess the subjective change in patients in relation to improvement in symptoms through the Subjective Global Scale | 7 days
  Assess the improvement in symptoms measured as the proportion of patients who present a change in the Global Subjective Scale during the 7 days after starting treatment with respect to the baseline measurement.
  The subjective global scale for symptom improvement compares with the score of the previous day to determine health status daily. Is consists of 1 question related to the progress in the symptoms presentation, the answers go from much better to really worse.
Assess the improvement in health status through the modified Likert Scale | 7 days
  To compare improvement in health status as a difference in the modified Likert scale by treatment group during the 7 days after starting treatment with respect to the baseline measurement.The patient will answer the scale daily.
  The Likert Scale is a seven point scale that is used to allow an individual to express how much they agree or disagree with a particular statement. The scale consists of 1 question associated to the health status of the patient. The possible answers go from Not feeling sick to feeling to Severely sick.

OTHER OUTCOMES:
Assess the percentage of patients with febrile episodes (≥38°C) during the intervention | 7 days
  The patient will report the presence of fever during the intervention, quantified with a thermometer.
To report the percentage of therapeutic adherence at day 7 of intervention by group of treatment | 7 days
  Adherence to treatment will be defined as a consumption ≥ 80% of the doses that the patient should have ingested at the time of the corresponding evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ana Luara Flores-Barranco, MD, Principal Investigator — Oaxaca Site Management Organization; Juan A Becerra-Hernández, MD, Principal Investigator — Centro de Investigación y Avances Médicos Especializados; Salvador Perez-Jaime, MD, Principal Investigator — CIMA; Victor C Bohorquez-Lopez, MD, Principal Investigator — Mérida Investigación Clínica
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heikkinen T, Jarvinen A. The common cold. Lancet. 2003 Jan 4;361(9351):51-9. doi: 10.1016/S0140-6736(03)12162-9. PMID 12517470
- [Background] Gonzales R, Malone DC, Maselli JH, Sande MA. Excessive antibiotic use for acute respiratory infections in the United States. Clin Infect Dis. 2001 Sep 15;33(6):757-62. doi: 10.1086/322627. Epub 2001 Aug 21. PMID 11512079
- [Background] Kirkpatrick GL. The common cold. Prim Care. 1996 Dec;23(4):657-75. doi: 10.1016/s0095-4543(05)70355-9. PMID 8890137
- [Background] Fendrick AM, Monto AS, Nightengale B, Sarnes M. The economic burden of non-influenza-related viral respiratory tract infection in the United States. Arch Intern Med. 2003 Feb 24;163(4):487-94. doi: 10.1001/archinte.163.4.487. PMID 12588210
- [Background] Passioti M, Maggina P, Megremis S, Papadopoulos NG. The common cold: potential for future prevention or cure. Curr Allergy Asthma Rep. 2014 Feb;14(2):413. doi: 10.1007/s11882-013-0413-5. PMID 24415465
- [Background] Dick EC, Jennings LC, Mink KA, Wartgow CD, Inhorn SL. Aerosol transmission of rhinovirus colds. J Infect Dis. 1987 Sep;156(3):442-8. doi: 10.1093/infdis/156.3.442. PMID 3039011
- [Background] Shaw Stewart PD. Seasonality and selective trends in viral acute respiratory tract infections. Med Hypotheses. 2016 Jan;86:104-19. doi: 10.1016/j.mehy.2015.11.005. Epub 2015 Nov 6. PMID 26608252
- [Background] Monto AS. Studies of the community and family: acute respiratory illness and infection. Epidemiol Rev. 1994;16(2):351-73. doi: 10.1093/oxfordjournals.epirev.a036158. PMID 7713184
- [Background] Lopez Olmedo N, Stern D, Perez Ferrer C, Gonzalez Morales R, Canto Osorio F, Barrientos Gutierrez T. Revision rapida: probabilidad de contagio por infecciones respiratorias agudas en el transporte publico colectivo. Salud Publica Mex. 2021 Feb 26;63(2, Mar-Abr):225-231. doi: 10.21149/12027. Spanish. PMID 33989481
- [Background] Nieman DC. Exercise, upper respiratory tract infection, and the immune system. Med Sci Sports Exerc. 1994 Feb;26(2):128-39. doi: 10.1249/00005768-199402000-00002. PMID 8164529
- [Background] Pitkaranta A, Nokso-Koivisto J, Jantti V, Takala A, Kilpi T, Hovi T. Lowered yields of virus-induced interferon production in leukocyte cultures and risk of recurrent respiratory infections in children. J Clin Virol. 1999 Dec;14(3):199-205. doi: 10.1016/s1386-6532(99)00056-6. PMID 10614857
- [Background] Turner RB. Epidemiology, pathogenesis, and treatment of the common cold. Ann Allergy Asthma Immunol. 1997 Jun;78(6):531-9; quiz 539-40. doi: 10.1016/S1081-1206(10)63213-9. PMID 9207716
- [Background] Eccles R. Understanding the symptoms of the common cold and influenza. Lancet Infect Dis. 2005 Nov;5(11):718-25. doi: 10.1016/S1473-3099(05)70270-X. PMID 16253889
- [Background] Douglas RG Jr, Alford RH, Cate TR, Couch RB. The leukocyte response during viral respiratory illness in man. Ann Intern Med. 1966 Mar;64(3):521-30. doi: 10.7326/0003-4819-64-3-521. No abstract available. PMID 4286006
- [Background] Hendley JO. Epidemiology, pathogenesis, and treatment of the common cold. Semin Pediatr Infect Dis. 1998 Jan;9(1):50-55. doi: 10.1016/S1045-1870(98)80051-4. Epub 2006 Jun 3. PMID 32288450
- [Background] Eccles R. Pathophysiology of nasal symptoms. Am J Rhinol. 2000 Sep-Oct;14(5):335-8. doi: 10.2500/105065800781329528. PMID 11068659
- [Background] Proud D, Reynolds CJ, Lacapra S, Kagey-Sobotka A, Lichtenstein LM, Naclerio RM. Nasal provocation with bradykinin induces symptoms of rhinitis and a sore throat. Am Rev Respir Dis. 1988 Mar;137(3):613-6. doi: 10.1164/ajrccm/137.3.613. PMID 3345041
- [Background] Conti B, Tabarean I, Andrei C, Bartfai T. Cytokines and fever. Front Biosci. 2004 May 1;9:1433-49. doi: 10.2741/1341. PMID 14977558
- [Background] Tyrrell DA, Cohen S, Schlarb JE. Signs and symptoms in common colds. Epidemiol Infect. 1993 Aug;111(1):143-56. doi: 10.1017/s0950268800056764. PMID 8394240
- [Background] JACKSON GG, DOWLING HF. Transmission of the common cold to volunteers under controlled conditions. IV. Specific immunity to the common cold. J Clin Invest. 1959 May;38(5):762-9. doi: 10.1172/JCI103857. No abstract available. PMID 13654511
- [Background] Macintyre S. Gender differences in the perceptions of common cold symptoms. Soc Sci Med. 1993 Jan;36(1):15-20. doi: 10.1016/0277-9536(93)90301-j. PMID 8424180
- [Background] Vos LM, Bruning AHL, Reitsma JB, Schuurman R, Riezebos-Brilman A, Hoepelman AIM, Oosterheert JJ. Rapid Molecular Tests for Influenza, Respiratory Syncytial Virus, and Other Respiratory Viruses: A Systematic Review of Diagnostic Accuracy and Clinical Impact Studies. Clin Infect Dis. 2019 Sep 13;69(7):1243-1253. doi: 10.1093/cid/ciz056. PMID 30689772
- [Background] Rhedin S, Lindstrand A, Rotzen-Ostlund M, Tolfvenstam T, Ohrmalm L, Rinder MR, Zweygberg-Wirgart B, Ortqvist A, Henriques-Normark B, Broliden K, Naucler P. Clinical utility of PCR for common viruses in acute respiratory illness. Pediatrics. 2014 Mar;133(3):e538-45. doi: 10.1542/peds.2013-3042. Epub 2014 Feb 24. PMID 24567027
- [Background] Barrett B, Locken K, Maberry R, Schwamman J, Brown R, Bobula J, Stauffacher EA. The Wisconsin Upper Respiratory Symptom Survey (WURSS): a new research instrument for assessing the common cold. J Fam Pract. 2002 Mar;51(3):265. PMID 11978238
- [Background] Barrett B, Brown R, Mundt M, Safdar N, Dye L, Maberry R, Alt J. The Wisconsin Upper Respiratory Symptom Survey is responsive, reliable, and valid. J Clin Epidemiol. 2005 Jun;58(6):609-17. doi: 10.1016/j.jclinepi.2004.11.019. PMID 15878475
- [Background] Barrett B, Brown RL, Mundt MP, Thomas GR, Barlow SK, Highstrom AD, Bahrainian M. Validation of a short form Wisconsin Upper Respiratory Symptom Survey (WURSS-21). Health Qual Life Outcomes. 2009 Aug 12;7:76. doi: 10.1186/1477-7525-7-76. PMID 19674476
- [Background] Lindberg F, Nelson I, Ranstam J, Riker DK. Early intervention with a glycerol throat spray containing cold-adapted cod trypsin after self-diagnosis of common cold: A randomised trial. PLoS One. 2022 Jul 5;17(7):e0270699. doi: 10.1371/journal.pone.0270699. eCollection 2022. PMID 35789217
- [Background] Eccles R, Winther B, Johnston SL, Robinson P, Trampisch M, Koelsch S. Efficacy and safety of iota-carrageenan nasal spray versus placebo in early treatment of the common cold in adults: the ICICC trial. Respir Res. 2015 Oct 5;16:121. doi: 10.1186/s12931-015-0281-8. PMID 26438038
- [Background] Barrett B, Brown R, Voland R, Maberry R, Turner R. Relations among questionnaire and laboratory measures of rhinovirus infection. Eur Respir J. 2006 Aug;28(2):358-63. doi: 10.1183/09031936.06.00002606. Epub 2006 Apr 26. PMID 16641127
- [Background] JACKSON GG, DOWLING HF, SPIESMAN IG, BOAND AV. Transmission of the common cold to volunteers under controlled conditions. I. The common cold as a clinical entity. AMA Arch Intern Med. 1958 Feb;101(2):267-78. doi: 10.1001/archinte.1958.00260140099015. No abstract available. PMID 13497324
- [Background] JACKSON GG, DOWLING HF, MULDOON RL. Acute respiratory diseases of viral etiology. VII. Present concepts of the common cold. Am J Public Health Nations Health. 1962 Jun;52(6):940-5. doi: 10.2105/ajph.52.6.940. No abstract available. PMID 14450587
- [Background] Hemila H. Vitamin C supplementation and common cold symptoms: problems with inaccurate reviews. Nutrition. 1996 Nov-Dec;12(11-12):804-9. doi: 10.1016/s0899-9007(96)00223-7. PMID 8974108
- [Background] West S, Brandon B, Stolley P, Rumrill R. A review of antihistamines and the common cold. Pediatrics. 1975 Jul;56(1):100-7. No abstract available. PMID 240145
- [Background] De Sutter AI, Saraswat A, van Driel ML. Antihistamines for the common cold. Cochrane Database Syst Rev. 2015 Nov 29;2015(11):CD009345. doi: 10.1002/14651858.CD009345.pub2. PMID 26615034
- [Background] Kim SY, Chang YJ, Cho HM, Hwang YW, Moon YS. Non-steroidal anti-inflammatory drugs for the common cold. Cochrane Database Syst Rev. 2015 Sep 21;2015(9):CD006362. doi: 10.1002/14651858.CD006362.pub4. PMID 26387658
- [Background] Eccles R. Efficacy and safety of over-the-counter analgesics in the treatment of common cold and flu. J Clin Pharm Ther. 2006 Aug;31(4):309-19. doi: 10.1111/j.1365-2710.2006.00754.x. PMID 16882099
- [Background] Handley DA, Magnetti A, Higgins AJ. Therapeutic advantages of third generation antihistamines. Expert Opin Investig Drugs. 1998 Jul;7(7):1045-54. doi: 10.1517/13543784.7.7.1045. PMID 15992014
- [Background] Clissold SP, Sorkin EM, Goa KL. Loratadine. A preliminary review of its pharmacodynamic properties and therapeutic efficacy. Drugs. 1989 Jan;37(1):42-57. doi: 10.2165/00003495-198937010-00003. PMID 2523301
- [Background] Kay GG, Harris AG. Loratadine: a non-sedating antihistamine. Review of its effects on cognition, psychomotor performance, mood and sedation. Clin Exp Allergy. 1999 Jul;29 Suppl 3:147-50. doi: 10.1046/j.1365-2222.1999.0290s3147.x. PMID 10444229
- [Background] Barenholtz HA, McLeod DC. Loratadine: a nonsedating antihistamine with once-daily dosing. DICP. 1989 Jun;23(6):445-50. doi: 10.1177/106002808902300601. PMID 2525847
- [Background] Haria M, Fitton A, Peters DH. Loratadine. A reappraisal of its pharmacological properties and therapeutic use in allergic disorders. Drugs. 1994 Oct;48(4):617-37. doi: 10.2165/00003495-199448040-00009. PMID 7528133
- [Background] Zhang J, Kan D. Evaluation of efficiency and safety of combined loratadine and budesonide in patients with anaphylactic rhinitis: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2022 Apr 29;101(17):e28851. doi: 10.1097/MD.0000000000028851. PMID 35512063
- [Background] Anolik R; Mometasone Furoate Nasal Spray With Loratadine Study Group. Clinical benefits of combination treatment with mometasone furoate nasal spray and loratadine vs monotherapy with mometasone furoate in the treatment of seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2008 Mar;100(3):264-71. doi: 10.1016/S1081-1206(10)60452-8. PMID 18426147
- [Background] Ratner PH, van Bavel JH, Martin BG, Hampel FC Jr, Howland WC 3rd, Rogenes PR, Westlund RE, Bowers BW, Cook CK. A comparison of the efficacy of fluticasone propionate aqueous nasal spray and loratadine, alone and in combination, for the treatment of seasonal allergic rhinitis. J Fam Pract. 1998 Aug;47(2):118-25. PMID 9722799
- [Background] Nayak AS, Philip G, Lu S, Malice MP, Reiss TF; Montelukast Fall Rhinitis Investigator Group. Efficacy and tolerability of montelukast alone or in combination with loratadine in seasonal allergic rhinitis: a multicenter, randomized, double-blind, placebo-controlled trial performed in the fall. Ann Allergy Asthma Immunol. 2002 Jun;88(6):592-600. doi: 10.1016/S1081-1206(10)61891-1. PMID 12086367
- [Background] Dahlen B, Roquet A, Inman MD, Karlsson O, Naya I, Anstren G, O'Byrne PM, Dahlen SE. Influence of zafirlukast and loratadine on exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2002 May;109(5):789-93. doi: 10.1067/mai.2002.123306. PMID 11994701
- [Background] Papi A, Papadopoulos NG, Stanciu LA, Degitz K, Holgate ST, Johnston SL. Effect of desloratadine and loratadine on rhinovirus-induced intercellular adhesion molecule 1 upregulation and promoter activation in respiratory epithelial cells. J Allergy Clin Immunol. 2001 Aug;108(2):221-8. doi: 10.1067/mai.2001.116861. PMID 11496238
- [Background] Berkowitz RB, Connell JT, Dietz AJ, Greenstein SM, Tinkelman DG. The effectiveness of the nonsedating antihistamine loratadine plus pseudoephedrine in the symptomatic management of the common cold. Ann Allergy. 1989 Oct;63(4):336-9. PMID 2529799
- [Background] Trukhan DI, Mazurov AL, Rechapova LA. [Acute respiratory viral infections: Topical issues of diagnosis, prevention and treatment in therapeutic practice]. Ter Arkh. 2016;88(11):76-82. doi: 10.17116/terarkh2016881176-82. Russian. PMID 28005035
- [Background] Chavez ML, DeKorte CJ. Valdecoxib: a review. Clin Ther. 2003 Mar;25(3):817-51. doi: 10.1016/s0149-2918(03)80110-8. PMID 12852704
- [Background] Wahbi AA, Hassan E, Hamdy D, Khamis E, Barary M. Spectrophotometric methods for the determination of Ibuprofen in tablets. Pak J Pharm Sci. 2005 Oct;18(4):1-6. PMID 16380350
- [Background] Potthast H, Dressman JB, Junginger HE, Midha KK, Oeser H, Shah VP, Vogelpoel H, Barends DM. Biowaiver monographs for immediate release solid oral dosage forms: ibuprofen. J Pharm Sci. 2005 Oct;94(10):2121-31. doi: 10.1002/jps.20444. PMID 16136567
- [Background] Varrassi G, Pergolizzi JV, Dowling P, Paladini A. Ibuprofen Safety at the Golden Anniversary: Are all NSAIDs the Same? A Narrative Review. Adv Ther. 2020 Jan;37(1):61-82. doi: 10.1007/s12325-019-01144-9. Epub 2019 Nov 8. PMID 31705437
- [Background] Bushra R, Aslam N. An overview of clinical pharmacology of Ibuprofen. Oman Med J. 2010 Jul;25(3):155-1661. doi: 10.5001/omj.2010.49. PMID 22043330
- [Background] Zoubek ME, Lucena MI, Andrade RJ, Stephens C. Systematic review: ibuprofen-induced liver injury. Aliment Pharmacol Ther. 2020 Mar;51(6):603-611. doi: 10.1111/apt.15645. Epub 2020 Jan 27. PMID 31984540
- [Background] Barkin RL. Acetaminophen, aspirin, or Ibuprofen in combination analgesic products. Am J Ther. 2001 Nov-Dec;8(6):433-42. doi: 10.1097/00045391-200111000-00008. PMID 11704782